CLINICAL TRIAL: NCT06516991
Title: Efficacy and Safety of Task-State-Based Temporal Interference Stimulation (TI) in Improving Depression in Patients With Bipolar Disorder
Brief Title: Task-State-Based Temporal Interference Stimulation (TI) to Improve Depression in Patients With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220008C-R2
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-07

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal Interference Stimulation (Experimental): Temporal Interference Stimulation
  Interventions: Device: Temporal Interference Stimulation

INTERVENTIONS:
Device: Temporal Interference Stimulation — Specific electrode sites are customized for the subject through magnetic resonance scanning, the deep nucleus cluster to be stimulated-nucleus accumbens is calibrated through electric field simulation before treatment, and the stimulation target can be accurately positioned by stimulating the specific electrode sites of the subject during treatment.
  During the treatment period, all subjects were treated with a fixed time interference stimulation (TI) device at a frequency of 30 minutes twice a day, 5 days a week, for a total of 10 treatments. The output current intensity during treatment is 3.64 mA+4.36 mA.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of temporal interference stimulation (TI) in improving depressive episodes of bipolar disorder, to analyze the therapeutic principle of TI in bipolar disorder depressive episodes based on task state MRI scanning, and to explore the abnormal regulation mechanism of anhedonia neural circuit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-50 years, right-handed, and completed nine years of compulsory education;
2. Meet the diagnostic criteria for bipolar disorder in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
3. HAMD-17: >17 points , assessed the presence of rapture deficits;
4. Subject had not been treated with a mood stabilizer, or had previously used an antidepressants and currently off medication for ≥1 week;
5. The subject/legal guardian is willing to actively cooperate with the treatment and sign an informed consent form after being fully informed of the temporal interference stimulus (TI).

Exclusion Criteria:

1. Co-morbid other psychiatric disorders, including affective psychiatric disorders, anxiety spectrum disorders, mental retardation, substance dependence (abuse), etc.;
2. History of a serious physical illness or a disease that may affect the central nervous system;
3. Neurologic disorders or risk of seizures such as previous cranial disorders, head trauma, abnormal electroencephalograms, magnetic resonance evidence of structural brain abnormalities, or a family history of epilepsy;
4. Contraindications to magnetic resonance scanning or time-interference stimulation (TI), such as the presence of metallic or electronic devices in the body (intracranial metallic foreign bodies, cochlear implants, pacemakers and stents, and other metallic foreign bodies);
5. Those who have received or are receiving electroconvulsive therapy (ECT ), modified electroconvulsive therapy (MECT ), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or other neurostimulation treatments;
6. Pregnant and lactating women, and women of childbearing age with positive urine pregnancy.

Ages: 16 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale（HAMD-17) | 0-5 days
  The Hamilton Depression Scale（HAMD-17) was used to assess the extent of the patient's depressive episodes, with higher scores representing more severe depression, and this scale was used to monitor the patient's improvement in depression before and after treatment.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale（MADRS） | 0-5 days
  The Montgomery-Asberg Depression Rating Scale (MADRS) is used to reflect the effectiveness of antidepressant treatment and to monitor changes in a patient's condition. The scale is a stand-alone scale whose ratings are based on a clinical interview with questioning about symptoms that leads to a rating of depression severity.
Hamilton Anxiety Scale（HAMA） | 0-5 days
  The Hamilton Anxiety Scale is primarily used for the assessment of anxiety levels, and has 14 items, each of which has a 0-4 scale, with anxiety possible above a score of 7. The higher the score, the more severe the anxiety.
Young Mania Rating Scale（YMRS） | 0-5 days
  The Young Mania Rating Scale is mainly used to assess the manic symptoms of the subjects before and after the treatment, there are 11 items, each symptom has a working scale, divided into 5 levels, the level score of each item is different, most of them are 0-4, in which the 5th, 6th, 8th and 9th items are scored as 0, 2, 4, 6, 8, and the higher the total score of the subject the more serious the degree of mania.
Snaith-Hamilton Pleasure Scale（SHAPS） | 0-5 days
  The Snaith-Hamilton Pleasure Scale is a self-report scale that assesses the degree of the subject's pleasure deficit; the higher the score, the more severe their pleasure deficit. The scale was used to assess the degree of improvement in the patients' pleasure deficit before and after treatment.
Temporal Experience of Pleasure Scale (TEPS) | 0-5 days
  The Temporal Experience of Pleasure Scale (TEPS) is a self-report scale that assesses an individual's anticipation and experience of future pleasure, with higher scores suggesting a stronger experience of pleasure. The scale was used to evaluate the degree of improvement of pleasure deficit before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Arm and interventions can be shared, while the clinical data will not be shared